CLINICAL TRIAL: NCT05597865
Title: Assessing the Feasibility of Economic Approaches to Prevent Substance Abuse Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21AA030225-01 (NIH); 1R21AA030225-01 (NIH)
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Adolescent Drinking; HIV/AIDS; Drug Use
MeSH Terms: conditions — Underage Drinking; Acquired Immunodeficiency Syndrome | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Other): Control arm will received Alcohol and Drug Use Risk Reduction Sessions
  Interventions: Behavioral: Alcohol and Drug Use Risk Reduction Sessions
- Intervention (Experimental): Participants in the intervention arm will receive four (4) Financial Literacy (FL) training sessions and receive a Youth Development Savings account (YDA) at a financial institution accredited by the Bank of Uganda for long-term savings. Each YDA account will be opened in the name of the participant. Savings will be matched at a 1:1 rate with money from the program.
  Interventions: Behavioral: Economic Empowerment Intervention; Behavioral: Alcohol and Drug Use Risk Reduction Sessions

INTERVENTIONS:
Behavioral: Economic Empowerment Intervention — Economic Empowerment Intervention comprising Financial Literacy Sessions and Youth Development Accounts
  Arms: Intervention
Behavioral: Alcohol and Drug Use Risk Reduction Sessions — All participants in the control and treatment arm will receive Alcohol and Drug Use Risk Reduction sessions tailored for Adolescents and Youths Living with HIV.

SUMMARY:
The proposed study will test the impact of an economic empowerment intervention on reducing alcohol and drug use (ADU) among adolescents and youth living with HIV (AYLHIV) in poverty-impacted communities in Uganda. It focuses on improving understanding of multi-level context- specific risk and protective factors for ADU among AYLHIV.

DETAILED DESCRIPTION:
Adolescent alcohol and drug use (ADU) is a significant public health challenge in sub-Saharan Africa (SSA). About 41.6% of adolescents in SSA reported using at least one psychoactive agent, with alcohol being the most commonly used drug. Uganda, one of the poorest countries in SSA, has the second highest rate of per capita alcohol consumption in SSA (15.1 liters of pure alcohol vs regional average of 6.2 liters of pure alcohol) and one third of Ugandan adolescents have used alcohol in their lifetime, 22.5 million are current drinkers, and over 50% engage in heavy episodic drinking. These estimates reach even greater magnitudes in the country's fishing villages - a key vulnerable population- where ADU is normative. A few studies have assessed ADU among AYLHIV, yet AYLHIV are at higher risk for ADU, and ADU impedes adherence to antiretroviral therapy (ART) retention in care, and viral suppression. Several studies have examined the risk and resilience factors for ADU but few interventions targeting ADU have been tested in SSA. . The majority of ADU interventions have been implemented in school settings, which may exclude adolescents in fishing communities that have high rates of school dropout. Moreover, none has targeted risk factors such as poverty and mental health, which are rampant among AYLHIV and their families, undermine AYLHIV's coping skills and resources, and have been associated with increased risk for ADU among adolescents. Economic empowerment (EE) interventions have the potential to prevent ADU among AYLHIV by reducing poverty and its associated mental health impacts, and also bolstering AYLHIV and their families' resources to overcome the challenges associated with HIV. Given the lack of evidence-based culturally tailored interventions to prevent ADU in AYLHIV in low-income settings such as Uganda, this study proposes to: Aim 1a. Examine the prevalence and consequences of ADU in a sample of 200 AYLHIV (ages 18-24) seen at six (6) HIV clinics located in the fishing communities of southwestern Uganda. ADU will be measured using self-report and biological data (i.e. urine). Aim 1b. Using a mixed methods approach, identify the multi-level (individual, interpersonal, community and structural) factors associated with ADU among AYLHIV. Aim 2: Using a subset of the sample, explore the feasibility and short-term effects of a EE intervention on ADU among AYLHIV. Our intervention focuses on older adolescents and young adults in a high-risk environment (i.e. fishing communities) to elucidate the contextually relevant risk and resilience factors for ADU among AYLHIV undergoing social transitions. Additionally we innovatively target the most commonly occurring risk and resilience factors for ADU (i.e. poverty and mental health problems) through the EE that includes provision of youth development savings accounts, financial literacy sessions and ADU risk reduction sessions.

ELIGIBILITY:
Inclusion Criteria for AYLHIV:

1. male or female AYLHIV aged 15-24 years;
2. medically diagnosed with HIV and aware of their HIV status;
3. enrolled in care at one of the selected HIV clinics.
4. positive self-report or urine test for alcohol or drug use

Exclusion Criteria:

1. any AYLHIV with negative urine alcohol or drug use test and negative self-report for alcohol and drug use
2. anyone with a significant cognitive impairment that interferes with their understanding of the informed consent process, or is unable/unwilling to consent.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Brathwaite, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- International Center for Child Health and Development Field Office, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available to other researchers through the NIH central data repositories upon request from the researcher. The researcher will be required to provide a research question, hypothesis, and analysis plan and strategies for maintaining data integrity in order to access the data.
Supporting Information: Study Protocol
Time Frame: These data will be available within 24 months after completing the study, and access will be maintained for 10 years.

REFERENCES:
- [Derived] Brathwaite R, Mutumba M, Nanteza J, Filiatreau LM, Migadde H, Namatovu P, Nabisere B, Mugisha J, Mwebembezi A, Ssewamala FM. Assessing the Feasibility of Economic Approaches to Prevent Substance Abuse Among Adolescents: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2023 Jun 14;12:e46486. doi: 10.2196/46486. PMID 37314844

RESULTS

PARTICIPANT FLOW:
Groups:
- Alcohol and Drug Use Risk Reduction Arm: Participants in the ADURR condition participated in four Alcohol and drug use risk reduction (ADURR) sessions focused on identifying and making decisions that align with values, managing individual risk-taking behaviors and peer pressure, strengthening interpersonal relationships, and goal setting.
- Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm: In addition to the adapted ADU training module that the ADURR-only group will receive, AYLHIV in the intervention arm will receive four (4) Financial Literacy Training (FLT) sessions and a Youth Development Savings account (YDA) for long-term savings. For the proposed study, the EE intervention will be in the form of a YDA, where savings are housed at a local bank and deposits made by the adolescent are matched by the intervention to encourage savings. Each AYLHIV in the EE intervention will receive a YDA held in their own name in a bank registered by the Central Bank (Bank of Uganda). We will form partnerships with national banks operating in the study area. The account will then be matched with money from the program. The maximum adolescent's contribution to be matched by the program will be an equivalent of US $20 per month per adolescent or US $120 for the 6-month intervention period.
Period: Overall Study
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Started | 46 | 49
Completed | 44 | 46
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm | Total
Number analyzed (Participants) | 46 | 49 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (2.21) | 22.0 (1.90) | 21.9 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 14 | 18 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 49 | 95
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Completing the Study at 6 Months
Description: Percentage of participants completing the study at 6 months
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 46 | 49
Participants | 44 | 46

2. Primary Outcome: Number of Participants Enrolling in the Study at Baseline
Description: Number of participants enrolling in the study at baseline
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 44 | 46
Participants | 44 | 46

3. Secondary Outcome: Percentage of Participants That Self-reported Use of Any Drug in the Last 3 Months at the Baseline Assessment
Description: Percentage of participants that self-reported use of any drug in last 3 months at the baseline assessment . Any of the drugs in the list of substances specified in the NIDA-Modified ASSIST questionnaire.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 46 | 49
Participants | 25 | 31

4. Secondary Outcome: Percentage of Participants That Self-reported Use of Any Drug in Last 3 Months at the 6-month Assessment
Description: Percentage of participants that self-reported use of any drug in last 3 months at the 6-month assessment. Any of the drugs in the list of substances specified in the NIDA-Modified ASSIST questionnaire.
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 44 | 46
Participants | 21 | 24

5. Secondary Outcome: Optimism Scale Total Score at Baseline
Description: Optimism scale measures hope that something good is going to happen in the future. Total score ranges from 9 to 45. Items were rated on a 5-item scale with higher scores are indicative of higher levels of optimism.
Time Frame: Baseline
Population: Score from Optimism scale
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 46 | 49
score | 38.5 (5.7) | 38.8 (5.4)

6. Secondary Outcome: Optimism Scale Total Score at 6 Months
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 44 | 46
score | 39.5 (4.4) | 39.3 (4.8)

7. Secondary Outcome: Beck Hopelessness Scale Total Score at Baseline
Description: Beck Hopelessness Scale total score at baseline is a 20-item scale that assesses negative expectations about the future. The total score ranges from 0-20. Higher scores indicate greater levels of hopelessness (more negative expectations about the future, less motivation, more pessimism.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 46 | 49
score | 4.6 (2.2) | 5.2 (3.0)

8. Secondary Outcome: Beck Hopelessness Scale Total Score at 6 Months
Description: as for outcome 7
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 44 | 46
score | 5.2 (3.0) | 4.4 (2.4)

9. Secondary Outcome: Depressive Symptoms Total Score at Baseline
Description: Center for Epidemiological Studies Depression Scale (CES-D). Total score range from 0-60. Higher scores indicate greater severity of depressive symptoms.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 46 | 49
score | 38.1 (10.8) | 37.6 (9.5)

10. Secondary Outcome: Depressive Symptom Total Score at 6 Months
Description: as for outcome 9
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 44 | 46
score | 37.6 (9.2) | 37.1 (9.1)

11. Secondary Outcome: Percentage of Participants That Self-reported Use of Any Drug in Last 12 Months at the Baseline Assessment
Description: Percentage of participants that self-reported use of any drug in last 12 months at the baseline assessment. Any of the drugs in the list of substances specified in the NIDA-Modified ASSIST questionnaire.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 46 | 49
Participants | 34 | 39

12. Secondary Outcome: Percentage of Participants That Self-reported Use of Any Drug in Last 12 Months at 6 Month Assessment
Description: Percentage of participants that self-reported use of any drug in last 12 months at the 6-month assessment. Any of the drugs in the list of substances specified in the NIDA-Modified ASSIST questionnaire.
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 44 | 46
Participants | 32 | 28

13. Secondary Outcome: Percentage of Participants That Self-reported Use of Alcohol in Last 12 Months at Baseline
Description: Percentage of participants that self-reported use of alcohol in the last 12 months at the baseline assessment.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 46 | 49
Participants | 31 | 35

14. Secondary Outcome: Percentage of Participants That Self-reported Use of Alcohol in Last 12 Months at the 6-month Assessment
Description: Percentage of participants that self-reported use of alcohol in the last 12 months at the 6-month assessment.
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 44 | 46
Participants | 29 | 26

15. Secondary Outcome: Percentage of Participants With a Positive Urine Test for Any Drug at Baseline
Description: Percentage of participants with a positive urine test for any drug at the baseline assessment
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 46 | 49
Participants | 15 | 24

16. Secondary Outcome: Percentage of Participants With a Positive Urine Test for Any Drug at the 6-month Assessment
Description: Percentage of participants with a positive urine test for any drug at the 6-month assessment
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 44 | 46
Participants | 11 | 15

17. Secondary Outcome: Percentage of Participants With a Positive Urine Test for Alcohol at the Baseline Assessment
Description: Percentage of participants with a positive urine test for alcohol at the baseline assessment
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 46 | 49
Participants | 8 | 20

18. Secondary Outcome: Percentage of Participants With a Positive Urine Test for Alcohol at the 6-month Assessment
Description: Percentage of participants with a positive urine test for alcohol at the 6-month assessment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
Number analyzed (Participants) | 44 | 46
Participants | 8 | 12

ADVERSE EVENTS:
Time Frame: baseline to 6 months follow-up
Arm/Group | Alcohol and Drug Use Risk Reduction Arm | Alcohol and Drug Use Risk Reduction + Economic Empowerment (ADURR+EE) Arm
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/49
Other Adverse Events (participants affected / at risk) | 0/46 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT05597865/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT05597865/SAP_001.pdf